CLINICAL TRIAL: NCT06567366
Title: A Single-Center, Prospective Study Evaluating the Efficacy and Safety of CAR T-cell Therapy in Combination With Glofitamab in the Treatment of Relapsed/Refractory Large B-Cell Lymphoma With High-Risk Prognostic Factors
Brief Title: CAR T-cell Therapy in Combination With Glofitamab for Relapsed/Refractory Large B-Cell Lymphoma With High-Risk Prognostic Factors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Prof., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Glofit-CART
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Large B-cell Lymphoma
MeSH Terms: interventions — Immunotherapy, Adoptive; glofitamab; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T-cell therapy in combination with Glofitamab (Experimental): After undergoing leukapheresis, participants will receive treatment in the following procedure.
  Bridging Phase:
  All participants will receive two cycles of Glofitamab treatment. On Day 1 of Cycle 1, patients will receive 1000 mg of Obinutuzumab as pretreatment.
  CAR-T Treatment Phase:
  Participants will receive lymphodepletion therapy with the FLU/CY regimen on Day -5 through Day -3. Participants will receive the CAR T-cell infusion on Day 0.
  Consolidation Phase:
  Treatment based on the response assessment at Day 28 after CAR T-cell infusion: participants who attained complete response (CR) at Day 28 will not receive additional Glofitamab treatment, while those attained partial response (PR), stable disease (SD), or progressive disease (PD) will receive additional four cycles of Glofitamab.
  Interventions: Biological: CAR T-cell therapy; Drug: Glofitamab; Drug: Obinutuzumab

INTERVENTIONS:
Biological: CAR T-cell therapy — Participants will receive CAR T-cell therapy via infusion on Day 0 (given as per treatment guidelines). Prior to CAR T-cell Therapy, participants will begin receiving lymphodepleting chemotherapy on Days -5 through -3 (given as per treatment guidelines).
Drug: Glofitamab — Glofitamab is given intravenously at a dose of 2.5mg over 4 hours on Cycle 1 Day 8.
  Glofitamab is given intravenously at a dose of 10mg over 2 hours on Cycle 1 Day 15.
  Glofitamab is given intravenously at a dose of 30mg over 2 hours on Day 1 of Cycles 2-6 (as relevant).
Drug: Obinutuzumab — Obinutuzumab pre-treatment is given intravenously at a dose of 1g on Cycle 1 Day 1.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of CAR T-cell therapy in combination with glofitamab for the treatment of relapsed/refractory large B-cell lymphoma with high-risk prognostic factors.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed Informed Consent Form
* Histologically confirmed large B-cell lymphoma with CD19 and CD20 expression, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS); primary mediastinal large B-cell lymphoma (PMBCL); high-grade B-cell lymphoma (HGBL); and transformed follicular lymphoma
* Patients who have relapsed or are refractory to at least prior first-line therapy, including anthracycline-containing chemotherapy regimens and anti-CD20 monoclonal antibody therapy
* Patients must be willing to receive CAR-T and Glofitamab therapy and be deemed suitable for CAR-T and Glofitamab treatment by the investigator
* Presence of at least one high-risk prognostic factor: (1) extranodal involvement; (2) maximum tumor diameter > 4 cm; (3) TP53 mutation
* ECOG Performance Status of 0, 1, or 2
* Life expectancy ≥12 weeks
* Adequate hematologic function (unless due to underlying disease, such as extensive bone marrow involvement, or secondary to lymphoma-related splenomegaly as determined by the investigator, but transfusion of blood products is allowed) and adequate liver, renal, pulmonary, and cardiac function

Key Exclusion Criteria:

* Hypersensitivity to any study drug or excipient
* History of allogeneic stem cell transplantation
* Patients with active viral hepatitis requiring treatment as determined by the investigator: chronic hepatitis B virus carriers with HBV DNA ≥ 500 IU/mL (2500 copies/mL) (HBV DNA testing only for patients who test positive for hepatitis B surface antigen or core antibody); patients who test positive for HCV RNA (HCV testing only for patients who test positive for HCV antibody)
* Presence of uncontrolled infection, cardio-cerebrovascular disease, coagulopathy, or autoimmune disease, etc
* History of HIV infection
* Presence or concurrence of other malignancies within the past 2 years, with the exception of cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors
* Previous anti-CD19 CAR-T therapy is not allowed
* Pregnant or lactating women
* Other uncontrollable medical condition that may interfere the participation of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | Up to 2 years
  CR rate is defined as the percentage of participants achieving CR per the Lugano Classification as determined by study investigators

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of participants achieving either CR or partial response (PR) per the Lugano Classification as determined by study investigators
Duration of Response (DoR) | Up to 2 years
  DoR is defined only for participants who experience an objective response and is the time from the first objective response to disease progression or death from any cause.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from leukapheresis to first documented progression or death from any cause.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from leukapheresis to death from any cause.
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 2 years
  Assessed by CTCAE criteria v5 and ASTCT 2019 criteria for CRS/ICANS adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China